CLINICAL TRIAL: NCT03391063
Title: Evaluation Of Chewing Efficiency Of Metal-Reinforced PolyAmide Denture Base In Comparison To Conventional Heat Cured Acrylic Resin Denture Base For Mandibular Complete Denture (A Randomized Clinical Trial)
Brief Title: Evaluation of Chewing Efficiency of Conventional Complete Denture in Comparison to Reinforced Poly Amide Denture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdallah Abdelmottaleb, dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Reinforced complete denture
Record Dates: First submitted 2017-12-29; First posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Mouth, Edentulous
MeSH Terms: conditions — Mouth, Edentulous | interventions — Nylons

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- reinforced polyamide denture base (Experimental): metal reinforced polyamide denture base
  Interventions: Other: polyamide
- conventional acrylic resin denture base (Active Comparator): conventional heat cured acrylic resin denture base
  Interventions: Other: heat cured acrylic resin

INTERVENTIONS:
Other: polyamide — metal reinforced polyamide denture base material
  Other Names: nylon
  Arms: reinforced polyamide denture base
Other: heat cured acrylic resin — conventional heat cured acrylic resin denture base material
  Arms: conventional acrylic resin denture base

SUMMARY:
the trial is done in order to reinforce polyamide to improve its modulus of elasticity to be able to use it as a denture base material in all clinical cases

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient with age range (45-55) completely edentulous and in good medical condition.
2. All patients have skeletal Angle's class I maxillo-mandibular relationship and have sufficient interarch distance.
3. Free from any systemic or neuromuscular disorder that might affect chewing efficiency of masticatory muscles.
4. Free from any tempro-mandibular joint disorder.
5. The patients have good oral hygiene.
6. The edentulous ridges should be covered by firm healthy mucosa.
7. Healthy and co-operative patients.

Exclusion Criteria:

1. Patients with bad habits as severe clenching or bruxism, drug or alcohol addiction, moderate or heavy smoking (greater than 10 cigarettes per day).
2. Previous history of radiotherapy or chemotherapy.
3. Any skeletal problem dictates surgical intervention.
4. Patients having hormonal disorders as diabetes, thyroid or parathyroid hormonal diseases were not included.
5. Patient with xerostomia or excessive salivation.
6. No intraoral soft and hard tissue pathosis.
7. Psychiatric problems.

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2018-05-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
chewing efficiency assessed using sieving method | 6 weeks
  chewing efficiency of the mandibular complete denture

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vojdani M, Giti R. Polyamide as a Denture Base Material: A Literature Review. J Dent (Shiraz). 2015 Mar;16(1 Suppl):1-9. PMID 26106628